CLINICAL TRIAL: NCT03858504
Title: The Comparison of the Effects of Yoga and Home Exercise Program in Children With Enthesitis Related Arthritis
Brief Title: Yoga Versus Home Exercise Program in Children With Enthesitis Related Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Collaborators: Dokuz Eylul University (Other); Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ezgi Yaşar, PT., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YOGAERA
Record Dates: First submitted 2019-02-27; First posted 2019-02-28 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Enthesitis Related Arthritis
Keywords: yoga; home exercises; juvenile idiopathic arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): The yoga program will include breathing exercises, different postures, and meditation. The yoga will be performed in groups. The program will be supervised a physical therapist for two times in a week for eight weeks . A session will be fifty minutes (5-10 minutes: warming-up, 20-25 minutes: postures, 10-15 minutes: cooling down).
  Interventions: Other: Exercise
- Home Exercise Group (Active Comparator): Home exercise program will consist of trunk strengthening exercises. The patients will be asked to check the exercise days. Patients will be contacted with telephone once a week.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The children with enthesitis related arthritis will be randomized into one of the exercise groups as yoga or home exercises and will perform the exercise program for 2 times a week for 8 weeks according to their groups.

SUMMARY:
The aim of this study is to compare the effectiveness of different exercises programs as 'Yoga' and 'Home Exercise' in Enthesitis Related Arthritis.

DETAILED DESCRIPTION:
Enthesitis is the localized inflammation in the attachments of muscles, ligaments, fascia to bone. Enthesitis related arthritis is a sub-form of Juvenile Idiopathic Arthritis (JIA) and primarily lower extremities, spine, and sacroiliac joints. In the literature, exercise therapy is found beneficial to improve bone density, muscle strength and functionality without leading adverse effects in these children.

Recently yoga has emerged as a new exercise approach which consist of both physical an mental components to improve self-awareness and mindfulness. However, the effects of yoga did not investigated in JIA patients. The only evidence is a case study which reports improvements in pain and stiffness in a child with JIA.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 13-18 years
2. Having a diagnosis of enthesitis related arthritis
3. Having a diagnosis at least 6 months ago
4. Being able to understand exercise instructions
5. Consent of family and the patient

Exclusion Criteria:

1. Any contraindication to perform exercise (neurological, cardiovascular etc.)
2. Change in medication

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in 6 minute walking distance | At baseline and 8 weeks later
  Six minute walking distance will be used for determining the functional status of lower extremity. The test will be performed in a 15-m corridor. The patient will be asked to walk as fast as possible without running. Standard instructions will be used for motivation. The patients will be allowed to stop if they want without stopping the chronometer. The total distance will be measured at the end of six minutes.
Change in timed up and down stair test | At baseline and 8 weeks later
  The patients will be asked to climb and descend 13 steps and the time will be recorded.

SECONDARY OUTCOMES:
Change in Quality of Life | At baseline and 8 weeks later
  Pediatric Quality of Life (PedsQL) 3.0 Arthritis Module will be used to assess the quality of life of the patients and their parents.It is a 22-item measure consisting of 5 scales: pain and hurt, daily activities, treatment, worry, and communication. Items are rated on a 5-point Likert scale (0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Often, 4 = Almost Always). The possible range of scores is 0-88 by summing subscale scores and lower scores indicates better quality of life.
Change in Pain | At baseline and 8 weeks later
  Numeric Rating Pain Scale will be used to assess pain severity. It has 11 points (0-10) where 0 represents no pain and 10 represents extreme pain.

CONTACTS AND LOCATIONS:
Overall Officials: Erdogan Kavlak, PhD, Study Director — Pamukkale University
Locations (1):
- Dokuz Eylul University, Faculty of Medicine, Nevvar Salih Isgoren Children's Hospital, Division of Pediatric Rheumatology, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henderson CJ, Lovell DJ, Specker BL, Campaigne BN. Physical activity in children with juvenile rheumatoid arthritis: quantification and evaluation. Arthritis Care Res. 1995 Jun;8(2):114-9. doi: 10.1002/art.1790080210. PMID 7794985
- [Background] Kirchheimer JC, Wanivenhaus A, Engel A. Does sport negatively influence joint scores in patients with juvenile rheumatoid arthritis. An 8-year prospective study. Rheumatol Int. 1993;12(6):239-42. doi: 10.1007/BF00301009. PMID 8484096
- [Background] Bacon MC, Nicholson C, Binder H, White PH. Juvenile rheumatoid arthritis. Aquatic exercise and lower-extremity function. Arthritis Care Res. 1991 Jun;4(2):102-5. doi: 10.1002/art.1790040207. PMID 11188589
- [Background] Tarakci E, Yeldan I, Baydogan SN, Olgar S, Kasapcopur O. Efficacy of a land-based home exercise programme for patients with juvenile idiopathic arthritis: a randomized, controlled, single-blind study. J Rehabil Med. 2012 Nov;44(11):962-7. doi: 10.2340/16501977-1051. PMID 23027068
- [Background] Kuntze G, Nesbitt C, Whittaker JL, Nettel-Aguirre A, Toomey C, Esau S, Doyle-Baker PK, Shank J, Brooks J, Benseler S, Emery CA. Exercise Therapy in Juvenile Idiopathic Arthritis: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2018 Jan;99(1):178-193.e1. doi: 10.1016/j.apmr.2017.05.030. Epub 2017 Jul 18. PMID 28729171
- [Background] Feinstein AB, Cohen LL, Masuda A, Griffin AT, Gamwell KL, Stiles MT, Angeles-Han ST, Prahalad S. Yoga Intervention for an Adolescent With Juvenile Idiopathic Arthritis: A Case Study. Adv Mind Body Med. 2018 Winter;32(1):13-20. PMID 29406303
- [Background] Haaz S, Bartlett SJ. Yoga for arthritis: a scoping review. Rheum Dis Clin North Am. 2011 Feb;37(1):33-46. doi: 10.1016/j.rdc.2010.11.001. Epub 2010 Dec 3. PMID 21220084
- [Background] Ebnezar J, Nagarathna R, Yogitha B, Nagendra HR. Effects of an integrated approach of hatha yoga therapy on functional disability, pain, and flexibility in osteoarthritis of the knee joint: a randomized controlled study. J Altern Complement Med. 2012 May;18(5):463-72. doi: 10.1089/acm.2010.0320. Epub 2012 Apr 26. PMID 22537508
- [Background] Jensen MP, McFarland CA. Increasing the reliability and validity of pain intensity measurement in chronic pain patients. Pain. 1993 Nov;55(2):195-203. doi: 10.1016/0304-3959(93)90148-I. PMID 8309709
- [Background] Lelieveld OT, Takken T, van der Net J, van Weert E. Validity of the 6-minute walking test in juvenile idiopathic arthritis. Arthritis Rheum. 2005 Apr 15;53(2):304-7. doi: 10.1002/art.21086. No abstract available. PMID 15818658
- [Background] Zaino CA, Marchese VG, Westcott SL. Timed up and down stairs test: preliminary reliability and validity of a new measure of functional mobility. Pediatr Phys Ther. 2004 Summer;16(2):90-8. doi: 10.1097/01.PEP.0000127564.08922.6A. PMID 17057533
- [Background] Tarakci E, Baydogan SN, Kasapcopur O, Dirican A. Cross-cultural adaptation, reliability, and validity of the Turkish version of PedsQL 3.0 Arthritis Module: a quality-of-life measure for patients with juvenile idiopathic arthritis in Turkey. Qual Life Res. 2013 Apr;22(3):531-6. doi: 10.1007/s11136-012-0180-0. Epub 2012 Apr 29. PMID 22544413
- [Background] Galantino ML, Galbavy R, Quinn L. Therapeutic effects of yoga for children: a systematic review of the literature. Pediatr Phys Ther. 2008 Spring;20(1):66-80. doi: 10.1097/PEP.0b013e31815f1208. PMID 18300936